CLINICAL TRIAL: NCT06416813
Title: Preventive Intervention Value of Drug-Coated Balloons in Vulnerable Coronary Atherosclerotic Plaques
Brief Title: Preventive Intervention Value of DCB in Vulnerable Coronary Atherosclerotic Plaques
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yong He (Other)
Responsible Party: Sponsor-Investigator, Yong He, Head of Cardiology, Professor, Chief Physician, Principal Investigator, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WestChinaH-CVD-005
Record Dates: First submitted 2024-05-02; First posted 2024-05-16 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GDMT (No Intervention)
- GDMT+DCB (Experimental)
  Interventions: Procedure: GDMT+DCB

INTERVENTIONS:
Procedure: GDMT+DCB — Preventive Intervention on Eligible Vulnerable Plaques Using DCB
  Arms: GDMT+DCB

SUMMARY:
The PASSIVATE-CAP study is an investigator-initiated, prospective, randomized, multicenter, open-label superiority trial focusing on acute coronary syndrome (ACS) patients with nonflow-limiting vulnerable plaques in nonculprit vessels. In this study, eligible patients were randomized at a 1:1 ratio into two groups: patients who received guideline-directed medical therapy (GDMT) and patients who received GDMT combined with a drug-coated balloon (DCB). In this study, the use of PCSK9 inhibitors was limited to inclisiran. The primary endpoint was the minimal lumen area of the target lesion 1 year after randomization. The secondary endpoints encompass a range of factors, including the proportion of patients with vulnerable plaques in the target vessel, fibrous cap thickness, lipid core arc of the target lesion, minimal lumen area of the target vessel, and extent of LDL-C reduction in patients treated with inclisiran.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Diagnosis of ACS with the intention to undergo ICA There exists a nonculprit lesion characterized by a single diameter stenosis greater than 50% in the major coronary artery segments (with diameters ranging from 2.75 to 4 mm).

QFR value > 0.8 The OCT examination suggests vulnerable plaques with a fibrous cap thickness of < 65 µm, along with at least two of the other three OCT criteria Minimum lumen area <3.5 mm² Lipid core angle >180° Presence of macrophages lesion length ≤30 mm Provide informed consent Life expectancy greater than 1 year

Exclusion Criteria:

Patients with three or more target lesions or with two target lesions in the same coronary artery left main stem lesions Ostial lesions Thrombotic lesions Severe calcification or angulated lesions True bifurcation lesions requiring stent implantation Advanced heart failure (NYHA III-IV) Ischemic stroke in the past 6 months or any history of cerebral hemorrhage at any time Severe valve disease or valve disease that may require surgical or percutaneous valve replacement Coronary artery anatomy obstructs the complete imaging of the segment of interest (including at least 5 mm beyond the narrow ends).

Diffuse coronary artery disease or the presence of ≥1 untreated nonculprit lesion (nonculprit blood flow-restricting lesion planned for staged PCI).

History of myocardial infarction, CABG, or PCI Coronary artery anatomy not suitable for PCI The potential comorbidity that may impact the completion of the trial process. The planned major surgery requires discontinuation of DAPT. History of PCSK9 inhibitor (such as evolocumab or alirocumab) use within 90 days prior to the first study visit.

Exposed to Inclisiran or any other non-PCSK9 monoclonal antibody targeted treatment within the 2 years preceding the initial study visit, whether as an investigational drug or a marketed medication.

History of allergy to the investigational drug, its excipients, or other siRNA drugs Females of childbearing potential, defined as all female subjects physiologically capable of becoming pregnant, unless they are using effective contraception during the administration of the investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Minimum luminal area | 1 year
  Minimum luminal cross-sectional area of the target lesion measured 1 year after randomization.

SECONDARY OUTCOMES:
proportion of patients with vulnerable plaques in the target vessel | 1 year
  proportion of patients with vulnerable plaques in the target vessel
fibrous cap thickness | 1 year
  Fibrous cap thickness
lipid core arc | 1 year
  The lipid core arc as visualized on optical coherence tomography (OCT) refers to the angular extent and characteristics of the lipid-rich region within an atherosclerotic plaque. On cross-sectional OCT imaging, the lipid core appears as an area with high backscattering and high signal attenuation, distinguishing it from the surrounding fibrous or calcified plaque components. The key features of the lipid core arc include the arc angle (the angular extent of the lipid core in degrees), the arc thickness (the maximal radial thickness of the lipid core), and the arc location (the position of the lipid core relative to the lumen and other plaque components).
Changes in LDL-C | 1 year
  The degree of changes in patients' LDL-C (low-density lipoprotein cholesterol) levels before and after treatment

OTHER OUTCOMES:
Target vessel failure | 1 year
  A composite endpoint event encompassing cardiac death, target vessel myocardial infarction, and ischemia-driven target vessel revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Sichuan Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Z, Zhang J, Zhou M, Liang S, Chen Y, Li C, Wang H, Wei J, Huang B, Wang M, He Y; PASSIVATE-CAP trial investigator. Rationale and Design of the PASSIVATE-CAP Trial: The Preventive Intervention Value of Drug-Coated Balloons in Vulnerable Coronary Atherosclerotic Plaques. Clin Cardiol. 2026 Jan;49(1):e70243. doi: 10.1002/clc.70243. PMID 41521574